CLINICAL TRIAL: NCT04874844
Title: Recombinant Anti-VEGFR2 Fully Human Monoclonal Antibody (JY025) Injection Combined With Gefitinib/Erlotinib as First-line Treatment Phase II and III Clinical Trials on the Efficacy and Safety of Patients With EGFR-mutant NSCLC
Brief Title: JY025 is a First-line Treatment for EGFR Mutated NSCLC Phase II and III Clinical Trials of Efficacy and Safety
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Dongfang Biotech Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFBT-JY025-NSCLC-2020-30I
Record Dates: First submitted 2021-04-12; First posted 2021-05-06 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: NSCLC
Keywords: Late or metastatic non-squamous non-small cells; EGFR mutations Patients; cell lung cancer.

STUDY DESIGN:
Intervention Model Description: Phase II single ;Phase III parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase II open label non-randomizedand ;Phase III randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test drug group (Other): Phase II Dose Addition Stage JY025 12MG / KG and 16mg / kg Q3W Givenate Combined EGFRTKI (Gifan Totibi 250mg or Erlotini 150mg) QD scheme, 6 cases of each dose group in group (Gifanibini 3 cases of Erlotini); 1 or 2 doses of JY025 in dose expansion phase Q3W administration combined with EGFR-TKI (50mg or Ellotini 150mg) QD scheme, each dose group 6 Examples of subjects (3 cases of Gifeng Tinib and Ellotini).
  Interventions: Biological: Recombinant anti-VEGFR2 fully human monoclonal antibody (JY025)
- Group type (Active Comparator): Phase III 396 patient JY025 injection and placebo combined with Notes Totibi / Erlotini (Gifeng Totibi 250mg or Erlotini 150mg) Q3W QD treatment group is randomly packet in 1: 1 ratio (in each group) Gifanibi and Erlotini are 2: 1)
  Interventions: Biological: Recombinant anti-VEGFR2 fully human monoclonal antibody (JY025)

INTERVENTIONS:
Biological: Recombinant anti-VEGFR2 fully human monoclonal antibody (JY025) — The ratio of subjects in the experimental drug group to the placebo control group is 1:1, and you will have a 50% probability of receiving JY025 combined with gefitinib or erlotinib, and a 50% probability of receiving placebo combined with gefitinib Or erlotinib.
  Blind people, researchers, nurses, research assistants, inspectors, applicants and blind statisticians involved in clinical trials.

SUMMARY:
The Phase II study is a multi-center, open, dose escalation and dose extension clinical trial. It is planned to enroll 24 patients; the phase III study is a multi-center, randomized, double-blind, placebo-controlled clinical trial. It is planned to enroll 396 patients, including patients with locally advanced or metastatic non-squamous non-small cell lung cancer with EGFR mutations (EGFR 19 exon deletion or 21 exon mutation).

DETAILED DESCRIPTION:
The Phase II study is a multi-center, open, dose escalation and dose extension clinical trial. It is planned to enroll 24 patients with locally advanced or metastatic non-squamous non-small cell lung cancer with EGFR mutation (EGFR 19 exon deletion or 21 exon mutation).

Dose escalation select JY025 12mg/kg and 16mg/kg Q3W administration combined with EGFRTKI (gefitinib 250mg or erlotinib 150mg) QD plan, each dose group enrolled 6 subjects, in the first cycle Perform DLT evaluation. If 2/6 cases or more of DLT occur at 12 mg/kg, then the extended phase dose is reduced to 10 mg/kg; if 16 mg/kg occurs at 2/6 cases or more of DLT, the extended phase test is not performed at this dose.

Dose expansion selects 1 or 2 doses of JY025 Q3W administration combined with EGFR-TKI (gefitinib 250mg or erlotinib 150mg) QD regimen, each dose group enrolled 6 subjects (gefitinib and Erlotinib (3 cases each).

The Phase III study is a multi-center, randomized, double-blind, placebo-controlled clinical trial. It is planned to enroll 396 patients with EGFR mutation (EGFR 19 exon deletion or 21 exon [L858R] mutation) with locally advanced or metastatic non-squamous non-small cell lung cancer.

The study included a test drug group and a placebo control group. The dosage regimen of the test drug group was: JY025 is based on phase II clinical recommended dose, once every 21 days, gefitinib 250mg or erlotinib 150mg once a day; placebo The dosage regimen of the control group is: placebo is based on phase II clinical recommended dose, once every 21 days, gefitinib 250mg or erlotinib 150mg once a day. The ratio of the test drug group to the placebo control group is 1:1, and they will receive continuous administration until confirmed disease progression, intolerable toxicity, or meet any of the criteria for stopping the study medication.

ELIGIBILITY:
Inclusion Criteria:

* (1) Fully understand the purpose of the experiment, the investigator judges that he can abide by the experiment protocol, and voluntarily sign a written informed consent.

  (2) The age at the time of signing the informed consent is ≥18 years old, regardless of gender.

  (3) Patients with non-squamous non-small cell lung cancer (NSCLC) diagnosed by histology/cytology.

  (4) According to the TNM staging of UICC 8th edition, it is determined as ⅢB (not suitable for surgery or radiotherapy)-IV stage NSCLC.

  (5) The patient has EGFR exon 19 deletion (19del) or 21 exon [L858R] mutation confirmed by the central laboratory (only tissue samples are accepted), and it is suitable for first-line treatment of EGFR-TKI.

  (6) Have not received any systemic treatment for non-small cell lung cancer in the past, and have not received any EGFR-TKI drug treatment. If the subject has received adjuvant/neo-adjuvant therapy and then relapses, but the end of adjuvant/neo-adjuvant therapy is more than 6 months after the first dose of this study, the subject can also be included in the group.

  (7) There is at least one measurable lesion based on RECISTv1.1. (8) The ECOG score is 0~1. (9) The functions of major organs and bone marrow are basically normal. It is required that no blood transfusion or hematopoietic stimulating factors have been used within 14 days before screening. The laboratory test results are the results within 7 days before the start of treatment:

  ①Cagulation function INR≤1.5×ULN, aPTT≤1.5×ULN (if the subject is receiving anticoagulant therapy Treatment, as long as the aPTT is within the expected treatment range of anticoagulant drugs);

  ②The subject's liver and kidney function meets the following conditions: total bilirubin≤1.5×ULN, ALT and AST≤2.5×ULN, if the liver is invaded by tumor, AST and ALT≤5×ULN; endogenous creatinine clearance ≥60mL/min (Cockcroft-Gault formula); urine protein is 0 or 1, or urine protein quantitative <1g/24h ；

  ③The blood routine meets: neutrophil count ≥1.5×109/L, platelet ≥100×109/L, hemoglobin ≥9g/dL.

  (10) Adverse reactions caused by previous local treatments, surgery or other anti-cancer treatments have recovered to ≤ CTCAE level 1 (except for hair loss).

  (11) The life expectancy of the patient is> 12 weeks. (12) Take effective contraceptive measures throughout the study period until 12 weeks after the last medication.

Exclusion Criteria:

1. The patient is positive for EGFR T790M mutation, positive for ALK fusion, or has any other co-mutations (a report is required if co-mutation has been tested, and testing is not mandatory if it has not been tested).
2. Suffered from other malignant tumors other than NSCLC within 5 years or at the same time (except cured skin basal cell carcinoma, prostate carcinoma in situ and cervical carcinoma in situ).
3. Symptomatic central nervous system (CNS) metastasis.
4. Received major surgery, needle biopsy or subcutaneous venous access device placement within 7 days before the start of study treatment. Any post-operative bleeding or wound complications occurred within 2 months before the start of study treatment.
5. Before the start of the study treatment, received radiotherapy in the bone marrow area ≥25% of the radiotherapy area, received palliative chest radiotherapy within 28 days, or received radiotherapy for local relief or prevention of symptoms (such as pain, bleeding or obstruction) within 7 days.
6. Idiopathic pulmonary fibrosis confirmed by CT/X-ray; X-ray confirmed or had acute lung injury,Pneumoconiosis; have or have had radiation pneumonia or drug-induced pneumonia; clinically active interstitial lung disease (chronic, stable,Except for asymptomatic patients with imaging changes); imaging evidence shows lung cavities.
7. Pleural effusion, pericardial effusion, or ascites and need to be drained every other week or more frequently.
8. Superior vena cava syndrome.
9. Patients with any serious and/or uncontrollable diseases, including:

   * Major cardiovascular disease (NYHA grade II-IV heart disease, myocardial infarction or under study Stroke occurred within 3 months before the start), unstable angina pectoris, unstable arrhythmia, congenital QT prolonged syndrome, or QTc interval corrected for the screening period> 500ms ( Bazetts formula: QTcB = QT/RR0.5); ②Past hypertensive crisis or history of hypertensive encephalopathy, hypertension not controlled by drugs (defined as systolic blood pressure ≥150mmHg and/or diastolic blood pressure >100mmHg);

     * Severe infections that are active or uncontrolled, such as nosocomial infections, bacteremia, severe lung infections, etc.; ④Patients with severe immunodeficiency (except those related to corticosteroid use), including those who are known to be HIV-positive; ⑤ Liver damage: Child-Pugh grade B (or worse) with severe liver cirrhosis; liver cirrhosis with a history of hepatic encephalopathy; clinically significant ascites caused by liver cirrhosis, which requires diuretic and/or puncture treatment; yes History of hepatorenal syndrome.
10. Evidence of major coagulopathy or other obvious bleeding tendency:

    * Bleeding incidents caused by esophageal and/or gastric varices occurred within 6 months before the start of the study treatment;

      * Hemoptysis occurred within 1 month before the start of study treatment (>2.5 mL bright red blood each time);

        * Thrombosis or embolism events, major vascular diseases (such as aortic aneurysms that require surgical repair) occurred within 6 months before the start of the study treatment; ④Current or recent (within 10 days before the start of the study treatment) anticoagulant therapy for therapeutic purposes (except for low molecular weight heparin therapy); ⑤Current or recent (within 10 days before the start of the study treatment) use aspirin (>325 mg/d) or ticlopidine, clopidogrel, cilostazol for treatment; ⑥Patients with imaging evidence that there are large blood vessels invaded or wrapped, and there is a significant risk of bleeding.
11. Abdominal or tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months before the start of study treatment.
12. Severe, non-healing or dehiscence wounds, active ulcers or untreated fractures.
13. There are factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea, and intestinal obstruction.
14. Being treated with CYP3A4 inducers (such as rifampicin or phenytoin) or strong inhibitors (such as itraconazole or ketoconazole).
15. Proton pump inhibitors (such as esomeprazole magnesium or omeprazole) need to be used daily.
16. Any known serious ocular surface disease.
17. Those who are known to be allergic to any component of the therapeutic drug, or have a history of allergy to monoclonal antibody therapy.
18. Previously received allogeneic stem cell or solid organ transplantation.
19. The research treatment was conducted within 4 weeks before the start of the research treatment.
20. Are pregnant or breastfeeding.
21. For any other disease, metabolic dysfunction, physical examination or clinical laboratory examination to find contraindications to the study drug, the investigator's judgment may affect the interpretation of the results, or may put the patient at a high risk of treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase II ：6-month progression-free survival rate | 6-month progression-free survival rate
  Progression-free survival (PFS) will statistically describe the lower quartile (Q1), median and upper quartile (Q3) and their corresponding 95% confidence intervals, and use the Kaplan-Meier method to fit Survival curve.
Phase III：BIRC-assessed at least 6 months progression-free survival (PFS) | BIRC-assessed at least 6 months progression-free survival (PFS)
  The progression-free survival ( PFS ) assessed by BIRC was statistically described by calculating the lower quartile ( Q1 ), median, upper quartile ( Q3 ) and their corresponding 95 % confidence interval. Hierarchical logrank test was used to compare the differences between groups, and Kaplan-Meier method was used to fit the survival curve. Stratified factors included EGFR mutation type ( 19del or L858R ), baseline tumor stage ( stage III or IV ), and brain metastasis ( yes or no ). HR and 95 % confidence interval were estimated by stratified COX proportional hazard model.

CONTACTS AND LOCATIONS:
Overall Officials: yuankai shi, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences